CLINICAL TRIAL: NCT02518295
Title: β-galactosidase Producing Probiotic Strains to Improve Lactose Digestion: Probiotic and Lactose Intolerance
Brief Title: β-galactosidase Producing Probiotic Strains to Improve Lactose Digestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 14.33. MET
Record Dates: First submitted 2015-07-16; First posted 2015-08-07 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Positive control (Active Comparator): Ultra high temperature (UHT) milk containing 18 g total lactose
  Interventions: Other: Positive control
- Positive control with S. thermophilus (Active Comparator): UHT milk containing 18 g total lactose+ S. thermophilus
  Interventions: Other: Probiotic S. thermophilus
- Positive control with B. longum (Active Comparator): UHT milk containing 18 g total lactose+ B. longum
  Interventions: Other: Probiotic B. longum
- Negative control (Placebo Comparator): Lactose free milk
  Interventions: Other: Negative control

INTERVENTIONS:
Other: Positive control — 200ml milk containing 18g lactose
  Arms: Positive control
Other: Probiotic S. thermophilus — 200ml milk containing 18g lactose + probiotic S. thermophilus
  Arms: Positive control with S. thermophilus
Other: Probiotic B. longum — 200ml milk containing 18g lactose + probiotic B. longum
  Arms: Positive control with B. longum
Other: Negative control — 200 ml of UHT Lactose free milk
  Arms: Negative control

SUMMARY:
The purpose of this study is to assess that two β-galactosidase Producing Probiotic Strains help improve lactose digestion in subjects with lactose maldigestion.

DETAILED DESCRIPTION:
The trial will be cross over, randomized in incomplete blocks, controlled, double-blind:

each subject will be administered 3 products out of 4 (positive control, probiotic Streptococcus (S.) thermophilus, probiotic Bifidobacterium (B.) longum, negative control) in a random order on 3 different days separated by a washout period of at least one week, and maximum 2 weeks between each challenge.

The total sample size is 42 enrolled subjects/37 completed Patients will be males and females aged between 20 and 65 years with positive hydrogen breath test.

ELIGIBILITY:
Inclusion Criteria:

1. HBT> delta 20ppm (compared with the baseline value) measured at screening visit before challenge tests
2. Having signed the informed consent or having provide his/her legal representative's informed consent

Exclusion Criteria:

1. Known Food allergy
2. Any obstructive (COPD, asthma…) or restrictive respiratory syndrome that may impact breath test measurements
3. Any medically relevant malabsorption syndrome
4. Any medically relevant chronic gut motility disorder other than Irritable Bowel Syndrome (IBS), assessed with Rome III questionnaire
5. Ongoing therapy with drugs known to affect gut motility
6. Any general antibiotherapy taken during or within 4 weeks of study onset
7. Use of lactase pill (eg. Lacdigest®), as well as yoghurt and probiotics, for at least 2 days prior to Visit 0b
8. Subject who cannot be expected to comply with the study procedures
9. Currently participating or having participated in another clinical trial during last 8 weeks prior to the beginning of this study.
10. To be a close collaborator to the Investigators, either in terms of Family relationship and/or professional relationship
11. Pregnancy, based on anamnesis

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Lactose malabsorption as represented by the increase of exhaled hydrogen compared to baseline measured by the hydrogen Breath Test (HBT) | HBT measured every hour during 4 hours after challenge (HBT curve)

SECONDARY OUTCOMES:
Assessment of improvement of lactose intolerance symptoms using a composite score equal to the sum of individual symptoms measured using a visual analog scale (VAS) | 4 hours after every milk intake, from the time of ingestion up to 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Duboux, Study Director — Société des Produits Nestlé (SPN); Gabriela Bergonzelli, PhD, Study Director — Société des Produits Nestlé (SPN)
Locations (1):
- Metabolic Unit, Lausanne, Switzerland